CLINICAL TRIAL: NCT00206531
Title: Role of Naive T-Cells in the Pathogenesis of T-Cell Decline and Long Term Persistence of HIV
Brief Title: The Role of Naive T-Cells in HIV Pathogenesis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Other Study IDs: 114/05
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-10-04 (Estimated); Status verified 2005-06

CONDITIONS: HIV Infections
Keywords: HIV-1; Naive T-cells; CD31; Treatment Naive
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
While HIV mainly infects mature T-cells it can also infect newly produced (or naïve) T-cells. These infected naïve T cells may then act a viral reservoir even in patients with undetectable viral loads. Understanding when and how these cells are infected is important because it could help us to understand why patients fail therapy even if they have a persistently undetectable viral load.

DETAILED DESCRIPTION:
The overall goal of this project is to provide a comprehensive analysis of the role of naïve T-cells in the pathogenesis of T-cell decline and long-term persistence of HIV infection.

The study is divided into two parts.

Part 1 aims to determine the origin of HIV infected naïve T-cells in vivo by assessing the viral relatedness between HIV strains from naïve and memory CD4 T-cells. To do this we will be studying ten chronically infected individuals. Naïve and memory CD4 T-cells from these individuals will be purified using a magnetic bead sorting (MACS) strategy. Envelope sequences will then be isolated and subjected to diversity calculation

Part 2 seeks to answer whether infection of naïve T-cells is established early in infection and what the effect of antiretroviral therapy is on this subset of T-cells. We will initially examine the relative proportion of CD31+ (recent thymic emigrants) and CD31- naive CD4+ T-cells in infected acute (n=15) and chronic (n=15) infection and uninfected (n=15) individuals compared with healthy controls. We will then prospectively test individuals prior to and at 3, 6, 12, 18 and 24 months following intiation of HAART (Highly Active Antiretroviral Therapy) in individuals with acute (n=10) and chronic (n=10) HIV infection. Immunophenotyping will detemine the proportion of naïve T-cells that are CD31+ and those that are CD31-. Naïve and memory T-cell subsets will again be purified and total and integrated HIV DNA will be quantified using real-time PCR.

ELIGIBILITY:
Inclusion Criteria:

-

Part 1:

- HIV positive by ELISA and Western Blot VL >2,000, CD4 >350

Part 2:

* HIV positive by ELISA and Western Blot
* Established Chronic infection (15 individuals)
* Acute infection (15 individuals).
* Any viral load or CD4 count.
* No therapy.
* Any individual who initiates HAART as determined by the treating physician

Exclusion Criteria:

* none

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75

CONTACTS AND LOCATIONS:
Overall Officials: Sharon R Lewin, Principal Investigator — Director, Infectious Diseases Unit, The Alfred Hospital; Jenny Hoy, Principal Investigator — Head Clinical Research Unit, Infectious Diseases Unit, Alfred Hospital
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia